CLINICAL TRIAL: NCT02604342
Title: Randomized, Multicenter, Phase III, Open-Label Study of Alectinib Versus Pemetrexed or Docetaxel in Anaplastic Lymphoma Kinase-Positive Advanced Non Small Cell Lung Cancer Patients Previously Treated With Platinum-Based Chemotherapy and Crizotinib
Brief Title: Alectinib Versus Pemetrexed or Docetaxel in Anaplastic Lymphoma Kinase (ALK)-Positive Advanced Non-Small Cell Lung Cancer (NSCLC) Participants Previously Treated With Platinum-Based Chemotherapy and Crizotinib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO29750; 2015-000634-29 (EudraCT Number)
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib; Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alectinib (Experimental): Participants will receive oral alectinib at a dose of 600 milligrams (mg) twice daily, taken with food until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Interventions: Drug: Alectinib
- Premetrexed/Docetaxel (Active Comparator): Participants will receive chemotherapy with either pemetrexed (500 milligrams per square meter [mg/m^2] of body surface area) or docetaxel (75 mg/m^2) intravenously.
  Interventions: Drug: Docetaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Alectinib — Participants will receive oral alectinib at a dose of 600 mg twice daily, taken with food until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Arms: Alectinib
Drug: Docetaxel — Participants will receive docetaxel at a dose of 75 mg/m^2 of body surface area intravenously every 3 weeks, until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Other Names: Taxotere®
  Arms: Premetrexed/Docetaxel
Drug: Pemetrexed — Participants will receive pemetrexed at a dose of 500 mg/m^2 of body surface area intravenously every 3 weeks, until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Other Names: Alimta®
  Arms: Premetrexed/Docetaxel

SUMMARY:
This randomized active-controlled multicenter Phase III open-label study will evaluate and compare between treatment groups the efficacy of alectinib versus chemotherapy in participants with ALK-positive advanced NSCLC who were previously treated with chemotherapy and crizotinib, as measured by investigator-assessed progression-free survival (PFS) and to evaluate and compare between treatment groups the central nervous system (CNS) objective response rate (C-ORR) in participants with measurable CNS metastases at baseline, as assessed by an Independent Review Committee (IRC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced or recurrent (Stage IIIB not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC that is ALK-positive. ALK positivity must have been determined by a validated fluorescence in situ hybridization (FISH) test (recommended probe, Vysis ALK Break-Apart Probe) or a validated immunohistochemistry (IHC) test (recommended antibody, clone D5F3)
* Participant had received two prior systemic lines of therapy, which must have included one line of platinum-based chemotherapy and one line of crizotinib
* Prior CNS or leptomeningeal metastases allowed if asymptomatic
* Participants with symptomatic CNS metastases for whom radiotherapy is not an option will be allowed to participate in this study
* Measurable disease by RECIST Version 1.1 prior to the administration of study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* For all females of childbearing potential, a negative pregnancy test must be obtained within 3 days before starting study treatment

Exclusion Criteria:

* Participants with a previous malignancy within the past 3 years are excluded (other than curatively treated basal cell carcinoma of the skin, early gastrointestinal [GI] cancer by endoscopic resection or in situ carcinoma of the cervix)
* Participants who have received any previous ALK inhibitor other than crizotinib
* Any GI disorder that may affect absorption of oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (54):
- Belgium (3):
  - GHdC Site Notre Dame, Charleroi
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
- MBAL Serdika EOOD, Sofia, Bulgaria
- France (7):
  - Centre Francois Baclesse, Caen
  - Hopital Bichat Claude Bernard ; Service de Pneumologie, Paris
  - Hopital Du Haut Leveque; Service Des Maladies Respiratoires, Pessac
  - Hopital Foch; Pneumologie, Suresnes
  - Hopital Sainte Musse; Pneumologie, Toulon
  - Hopital Larrey; Pneumologie, Toulouse
  - Hopital Robert Schuman; Pneumologie, Vantoux
- Germany (5):
  - Zentralklinik Bad Berka GmbH; Abteilung Onkologie und Hämatologie, Bad Berka
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Asklepios-Fachkliniken Muenchen-Gauting; Onkologie, Gauting
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Pius-Hospital; Klinik fuer Haematologie und Onkologie, Oldenburg
- Hong Kong (2):
  - Queen Elizabeth Hospital; Clinical Oncology, Hong Kong
  - Queen Mary Hospital; Dept. of Clinical Oncology, Hong Kong
- Semmelweis Egyetem X; Pulmonologiai Klinika, Budapest, Hungary
- Italy (10):
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialita San Giuseppe Moscati, Avellino, Campania
  - AORN Ospedali dei Colli Ospedale Monaldi; UOC Pneumologia ad indirizzo Oncologico, Napoli, Campania
  - Istituto Nazionale Tumori Fondazione G. Pascale; U.O.C. Oncologia Medica Toraco Polmonare, Napoli, Campania
  - Ospedale Provinciale Santa Maria Delle Croci; Oncologia Medica, Ravenna, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini; U.O.C. Pneumologia Ad Indirizzo Oncologico 1, Rome, Lazio
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - POLICLINICO RODOLICO, U.O. di Oncologia Medica, Catania, Sicily
  - A.O. Universitaria Pisana-Ospedale Cisanello; Dipartimento Cardio Toracico-Pneumologia Ii, Pisa, Tuscany
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; Oncologia Medica, Perugia, Umbria
- Oslo Universitetssykehus HF; Radiumhospitalet, Oslo, Norway
- Medical University of Gdansk, Gdansk, Poland
- Portugal (3):
  - Hospital Geral; Servico de Pneumologia, Coimbra
  - IPO do Porto; Servico de Oncologia Medica, Porto
  - CHVNG/E_Unidade 1; Servico de Pneumologia, Vila Nova de Gaia
- Russia (6):
  - University сlinic of headaches, Moscow, Moscow Oblast
  - FSBI"National Medical Research Center of Oncology named after N.N.Petrov" MHRF, Saint Petersburg, Sankt-Peterburg
  - Main Military Clinical Hospital named after N.N. Burdenko, Moscow
  - City Clinical Oncology Hospital, Moscow
  - City Clinical Oncology Dispensary, Saint Petersburg
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg
- Slovakia (2):
  - FNsP F. D. Roosevelta Banska Bystrica, II.Ocna klinika SZU, Banská Bystrica
  - Vychodoslovensky onkologicky ustav, Košice
- South Korea (2):
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Korea University Guro Hospital; Oncology, Seoul
- Spain (5):
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Turkey (Türkiye) (5):
  - Adana Acıbadem Hospital Oncology Department, Adana
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Ankara
  - Istanbul Uni Capa Medical Faculty; Inst. of Oncology, Istanbul
  - Ege University Medical Faculty; Chest Diseases, Izmir
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya

REFERENCES:
- [Derived] Sikkema BJ, Baart SJ, Paats MS, Smit EF, Schols AMWJ, Mathijssen RHJ, van Rossum EFC, Dingemans AC. Body Weight Gain Associated With Alectinib in Patients With ALK+ Non-Small Cell Lung Cancer: Pooled Analysis of Individual Patient Data From Four Prospective Clinical Trials. J Clin Oncol. 2025 Feb 20;43(6):641-650. doi: 10.1200/JCO-24-01579. Epub 2024 Dec 11. PMID 39661917
- [Derived] Novello S, Mazieres J, Oh IJ, de Castro J, Migliorino MR, Helland A, Dziadziuszko R, Griesinger F, Kotb A, Zeaiter A, Cardona A, Balas B, Johannsdottir HK, Das-Gupta A, Wolf J. Alectinib versus chemotherapy in crizotinib-pretreated anaplastic lymphoma kinase (ALK)-positive non-small-cell lung cancer: results from the phase III ALUR study. Ann Oncol. 2018 Jun 1;29(6):1409-1416. doi: 10.1093/annonc/mdy121. PMID 29668860

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited participants with Anaplastic Lymphoma Kinase (ALK)-positive advanced Non-Small Cell Lung Cancer (NSCLC) in 13 countries from November 2015 to March 2017.
Pre-assignment Details: A total of 119 participants were enrolled and randomized into the study: 79 participants in the alectinib arm, and 40 participants in the chemotherapy arm.
Groups:
- Experimental: Alectinib: Participants received oral alectinib at a dose of 600 milligrams (mg) twice daily, taken with food and treatment continued until disease progression, unacceptable toxicity, withdrawal of consent or death.
- Active Comparator: Premetrexed/Docetaxel: Participants received chemotherapy with either pemetrexed (500 milligrams per square meter [mg/m^2] of body surface area) or docetaxel (75 mg/m^2) intravenously.
Period: Overall Study
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Started | 79 | 40
Completed | 36 | 17
Not Completed | 43 | 23
Not completed — Death | 32 | 16
Not completed — Progression of disease | 1 | 0
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Other | 1 | 0
Not completed — Study Termination by Sponsor | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized in the study, irrespective of whether or not they received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel | Total
Number analyzed (Participants) | 79 | 40 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (13.0) | 58.8 (10.5) | 56.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 20 | 53
  Male | 46 | 20 | 66
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 68 | 34 | 102
  Not reported | 4 | 1 | 5
  Unknown | 0 | 1 | 1
  Missing | 2 | 0 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 67 | 32 | 99
  Asian | 6 | 8 | 14
  Unknown | 5 | 0 | 5
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigator
Description: PFS was defined as the time from randomization to the first documented disease progression, as determined using RECIST v1.1, or death from any cause, whichever occurred first. As per RECIST v1.1, disease progression is a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 millimeter (mm) and the appearance of new lesions.
Time Frame: Randomization to first documented disease progression, death from any cause, or study end (up to 33 months)
Population: ITT population included all participants randomized in the study, irrespective of whether or not they received study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
months | 10.9 [8.1 to 15.5] | 1.4 [1.2 to 1.6]
Statistical Analysis 1: Comparison: Experimental: Alectinib vs Active Comparator: Premetrexed/Docetaxel; Test type: Superiority; p < 0.001, Stratified log-rank test; Hazard Ratio (HR) = 0.20, 95% CI 2-sided [0.12 to 0.33] — Estimated hazard ratio obtained from stratified Cox model with treatment group as covariate

2. Secondary Outcome: Percentage of Participants With CNS Objective Response Rate (ORR) With Measurable CNS Metastases at Baseline Using RECIST Version 1.1 as Assessed By IRC
Description: Overall response rate in subjects with confirmed CNS response (C-ORR) was defined as the percentage of subjects who attained Complete Response (CR) or Partial Response (PR) for lesions in the CNS. As per RECIST v1.1, CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm, PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Baseline through study end (up to 33 months)
Population: ITT population with measurable CNS metastasis (mc-ITT) included all participants in ITT population with measurable CNS metastasis at baseline (as per IRC).
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 24 | 17
percentage of participants | 66.7 | 0.0
Statistical Analysis 1: Comparison: Experimental: Alectinib vs Active Comparator: Premetrexed/Docetaxel; 95% confidence interval of the difference (alectinib - chemotherapy) computed using Hauck-Anderson approach; Test type: Superiority; p < 0.001, Chi-squared; Difference in C-ORR = 0.667, 95% CI 2-sided [0.39 to 0.86]

3. Secondary Outcome: PFS Using RECIST Version 1.1 as Assessed by IRC
Description: PFS was defined as the time from randomization to the first documented disease progression, as determined using RECIST v1.1, or death from any cause, whichever occurred first. As per RECIST v1.1, disease progression is a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 mm and the appearance of new lesions.
  This outcome measure was assessed as part of the primary analysis and was not repeated during final analysis.
Time Frame: Approximately 15 months (Tumor assessments at baseline, every 6 weeks until progressive disease (PD), death or withdrawal from study prior to PD)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 72 | 35
months | 7.1 [6.3 to 10.8] | 1.6 [1.3 to 4.1]

4. Secondary Outcome: Percentage of Participants With Objective Response of CR or PR Using RECIST Version 1.1 as Assessed by Investigator and IRC
Description: ORR was defined as the percentage of participants who attained CR or PR. As per RECIST v1.1, CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm, PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
  The IRC assessment was part of the primary analysis and was not repeated during final analysis.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
percentage of participants
  Assessed by Investigator | 50.6 | 2.5
  Assessed by IRC: number analyzed (Participants) | 72 | 35
  Assessed by IRC | 36.1 | 11.4

5. Secondary Outcome: Percentage of Participants With Disease Control Using RECIST Version 1.1 as Assessed by Investigator and IRC
Description: Disease control rate (DCR) was defined as the percentage of participants who attained CR, PR, or stable disease (SD) of at least 5 weeks. As per RECIST v1.1, CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm, PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters, SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters since the treatment started.
  The IRC assessment was part of the primary analysis and was not repeated during final analysis.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
percentage of participants
  Assessed by Investigator | 86.1 | 25.0
  Assessed by IRC: number analyzed (Participants) | 72 | 35
  Assessed by IRC | 76.4 | 48.6

6. Secondary Outcome: Duration of Response (DOR) Using RECIST Version 1.1 as Assessed by Investigator and IRC
Description: DOR was defined as the time from when response (CR or PR) was first documented to first documented disease progression or death, whichever occurred first. DOR was evaluated for participants who had a best overall response (BOR) of CR or PR.
  The IRC assessment was part of the primary analysis and was not repeated during final analysis.
Time Frame: From the first documented CR or PR to the first documented disease progression, death, or study end (up to 33 months)
Population: ITT population included all participants randomized in the study, irrespective of whether or not they received study drug. Number analyzed indicates number of participants with a BOR of CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
months
  Assessed by Investigator: number analyzed (Participants) | 40 | 1
  Assessed by Investigator | 12.0 [8.3 to 23.5] | 2.7 [NA to NA] — CI could not be calculated due to insufficient number of participants with the event
  Assessed by IRC: number analyzed (Participants) | 26 | 4
  Assessed by IRC | 9.7 [5.6 to NA] — The upper CI limit could not be calculated due to an insufficient number of participants with the event | NA [NA to NA] — Values could not be calculated due to an insufficient number of participants with the event

7. Secondary Outcome: PFS in C-ITT Population Using RECIST Version 1.1 as Assessed by Investigator and IRC
Description: PFS was defined as the time from randomization to the first documented disease progression, as determined using RECIST v1.1, or death from any cause, whichever occurred first. As per RECIST v1.1, disease progression is a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 mm and the appearance of new lesions.
  This outcome measure assessment was part of the primary analysis and was not repeated during final analysis.
Time Frame: as for outcome 3
Population: Intent-to-treat population with CNS metastasis (C-ITT) included participants in ITT population with CNS metastasis at baseline (as per IRC assessment).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 50 | 26
months
  Assessed by Investigator | 9.7 [6.9 to NA] — The upper limit of CI was not reached due to less number of participants with the event. | 1.4 [1.2 to 1.6]
  Assessed by IRC | 8.1 [6.3 to NA] — The upper limit of CI was not reached due to less number of participants with the event. | 1.5 [1.2 to 4.1]

8. Secondary Outcome: Time to CNS Progression in C-ITT Population Using RECIST Version 1.1 as Assessed by IRC
Description: Time to CNS progression was defined as the time from randomization until radiographic evidence of CNS progression. As per RECIST v1.1, disease progression is a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 mm and the appearance of new lesions.
  This outcome measure assessment was part of the primary analysis and was not repeated during final analysis.
Time Frame: as for outcome 3
Population: C-ITT included participants in ITT population with CNS metastasis at baseline (as per IRC assessment).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 50 | 26
months | NA [6.8 to NA] — The median and upper limit of CI was not reached due to less number of participants with the event. | 1.6 [1.3 to 9.9]

9. Secondary Outcome: Percentage of Participants With Disease Control in C-ITT Population Using RECIST Version 1.1 as Assessed by IRC
Description: Disease Control Rate (DCR) was defined as the percentage of participants who attained CR, PR, or stable disease (SD) of at least 5 weeks. As per RECIST v1.1, CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm, PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters, SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters since the treatment started.
Time Frame: From first documented CR, PR, or SD lasting at least 5 weeks through study end (up to 33 months)
Population: C-ITT included participants in ITT population with CNS metastasis at baseline (as per IRC assessment).
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 52 | 28
percentage of participants | 82.7 | 25.0

10. Secondary Outcome: Percentage of Participants With ORR in C-ITT Population Using RECIST Version 1.1 as Assessed by IRC
Description: ORR was defined as the percentage of participants who attained CR or PR. As per RECIST v1.1, CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm, PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Baseline through study end (up to 33 months)
Population: C-ITT included participants in ITT population with CNS metastasis at baseline (as per IRC assessment).
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 52 | 28
percentage of participants | 48.1 | 0.0

11. Secondary Outcome: Duration of Response for Lesions in the CNS (C-DOR) Using RECIST Version 1.1 as Assessed by IRC
Description: DOR was defined as the time from when response (CR or PR) was first documented to first documented disease progression or death, whichever occurred first. C-DOR was defined in a similar way for lesions in the CNS, taking into account all lesions in the body. DOR was evaluated for participants who had a BOR of CR or PR.
Time Frame: From the first documented CR or PR to the first documented disease progression, death, or study end (up to 33 months)
Population: C-ITT included participants in ITT population with CNS metastasis at baseline (as per IRC assessment). Number analyzed indicates number of participants with a BOR of CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 52 | 28
months | 13.9 [6.2 to 13.9] | NA [NA to NA] — Could not be calculated due to insufficient number of participants with the event

12. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from randomization to death from any cause. OS was confounded by cross-over of participants to the alectinib arm.
Time Frame: Randomization to death from any cause, through study end (up to 33 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
months | 27.8 [18.2 to NA] — The upper limit of CI was not reached due to less number of participants with the event. | NA [8.6 to NA] — The median and CI was not reached due to less number of participants with the event.

13. Secondary Outcome: Plasma Concentration of Alectinib
Time Frame: Predose (2 hours) at Baseline, Week 3 and Week 6
Population: The Pharmacokinetic (PK) Evaluable Population included all participants who received any dose of alectinib and who had at least one post-baseline PK sample available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Experimental: Alectinib
Number analyzed (Participants) | 56
nanogram/milliliter (ng/mL) | 559 (48.0)

14. Secondary Outcome: Plasma Concentration of Alectinib Metabolite
Time Frame: Predose (2 hours) at Baseline, Week 3 and Week 6
Population: The PK Evaluable Population included all participants who received any dose of alectinib and who had at least one post-baseline PK sample available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Experimental: Alectinib
Number analyzed (Participants) | 56
ng/mL | 240 (44.8)

15. Secondary Outcome: Compliance of European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) Over Time
Description: Percentage of participants who filled out an EORTC QLQ-C30 questionnaire at a visit. The EORTC QLQ-C30 questionnaire consisted of 30 questions generating five functional scores (physical, role, cognitive, emotional, and social); a global health status/global quality of life scale score; three symptom scale scores (fatigue, pain, and nausea and vomiting); and six stand alone one-item scores that capture additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and perceived financial burden.
Time Frame: Baseline through Week 138
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
percentage of participants
  Baseline: number analyzed (Participants) | 73 | 34
  Baseline | 92.4 | 85.0
  Treatment - Week 3: number analyzed (Participants) | 73 | 30
  Treatment - Week 3 | 96.1 | 83.3
  Treatment - Week 6: number analyzed (Participants) | 70 | 18
  Treatment - Week 6 | 97.2 | 60.0
  Treatment - Week 12: number analyzed (Participants) | 64 | 8
  Treatment - Week 12 | 95.5 | 80.0
  Treatment - Week 18: number analyzed (Participants) | 54 | 4
  Treatment - Week 18 | 88.5 | 50.0
  Treatment - Week 24: number analyzed (Participants) | 51 | 3
  Treatment - Week 24 | 91.1 | 100
  Treatment - Week 30: number analyzed (Participants) | 51 | 2
  Treatment - Week 30 | 96.2 | 66.7
  Treatment - Week 36: number analyzed (Participants) | 44 | 2
  Treatment - Week 36 | 89.8 | 66.7
  Treatment - Week 42: number analyzed (Participants) | 41 | 2
  Treatment - Week 42 | 95.3 | 66.7
  Treatment - Week 48: number analyzed (Participants) | 37 | 2
  Treatment - Week 48 | 100 | 100
  Treatment - Week 54: number analyzed (Participants) | 34 | 2
  Treatment - Week 54 | 97.1 | 100
  Treatment - Week 60: number analyzed (Participants) | 29 | 2
  Treatment - Week 60 | 100 | 100
  Treatment - Week 66: number analyzed (Participants) | 26 | 2
  Treatment - Week 66 | 89.7 | 100
  Treatment - Week 72: number analyzed (Participants) | 24 | 2
  Treatment - Week 72 | 88.9 | 100
  Treatment - Week 78: number analyzed (Participants) | 22 | 0
  Treatment - Week 78 | 84.6 |
  Treatment - Week 84: number analyzed (Participants) | 18 | 0
  Treatment - Week 84 | 78.3 |
  Treatment - Week 90: number analyzed (Participants) | 16 | 0
  Treatment - Week 90 | 88.9 |
  Treatment - Week 96: number analyzed (Participants) | 15 | 0
  Treatment - Week 96 | 93.8 |
  Treatment - Week 102: number analyzed (Participants) | 11 | 0
  Treatment - Week 102 | 84.6 |
  Treatment - Week 108: number analyzed (Participants) | 10 | 0
  Treatment - Week 108 | 100 |
  Treatment - Week 114: number analyzed (Participants) | 5 | 0
  Treatment - Week 114 | 83.3 |
  Treatment - Week 120: number analyzed (Participants) | 5 | 0
  Treatment - Week 120 | 100 |
  Treatment - Week 126: number analyzed (Participants) | 3 | 0
  Treatment - Week 126 | 100 |
  Treatment - Week 132: number analyzed (Participants) | 1 | 0
  Treatment - Week 132 | 100 |
  Treatment - Week 138: number analyzed (Participants) | 1 | 0
  Treatment - Week 138 | 100 |

16. Secondary Outcome: Compliance of European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer-13 (EORTC QLQ-LC13) Over Time
Description: Percentage of participants who filled out an EORTC QLQ-LC13 questionnaire at a visit. The EORTC QLQ-LC13 module generated one multiple-item scale score assessing dyspnea and a series of single item scores assessing chest pain, arm/shoulder pain, pain in other parts, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis.
Time Frame: Baseline through Week 138
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
percentage of participants
  Baseline: number analyzed (Participants) | 73 | 33
  Baseline | 92.4 | 82.5
  Treatment - Week 3: number analyzed (Participants) | 73 | 30
  Treatment - Week 3 | 96.1 | 83.3
  Treatment - Week 6: number analyzed (Participants) | 70 | 19
  Treatment - Week 6 | 97.2 | 63.3
  Treatment - Week 12: number analyzed (Participants) | 64 | 8
  Treatment - Week 12 | 95.5 | 80.0
  Treatment - Week 18: number analyzed (Participants) | 54 | 4
  Treatment - Week 18 | 88.5 | 50.0
  Treatment - Week 24: number analyzed (Participants) | 51 | 3
  Treatment - Week 24 | 91.1 | 100
  Treatment - Week 30: number analyzed (Participants) | 51 | 2
  Treatment - Week 30 | 96.2 | 66.7
  Treatment - Week 36: number analyzed (Participants) | 43 | 2
  Treatment - Week 36 | 87.8 | 66.7
  Treatment - Week 42: number analyzed (Participants) | 41 | 2
  Treatment - Week 42 | 95.3 | 66.7
  Treatment - Week 48: number analyzed (Participants) | 37 | 2
  Treatment - Week 48 | 100 | 100
  Treatment - Week 54: number analyzed (Participants) | 34 | 2
  Treatment - Week 54 | 97.1 | 100
  Treatment - Week 60: number analyzed (Participants) | 29 | 2
  Treatment - Week 60 | 100 | 100
  Treatment - Week 66: number analyzed (Participants) | 26 | 2
  Treatment - Week 66 | 89.7 | 100
  Treatment - Week 72: number analyzed (Participants) | 24 | 2
  Treatment - Week 72 | 88.9 | 100
  Treatment - Week 78: number analyzed (Participants) | 22 | 0
  Treatment - Week 78 | 84.6 |
  Treatment - Week 84: number analyzed (Participants) | 18 | 0
  Treatment - Week 84 | 78.3 |
  Treatment - Week 90: number analyzed (Participants) | 16 | 0
  Treatment - Week 90 | 88.9 |
  Treatment - Week 96: number analyzed (Participants) | 16 | 0
  Treatment - Week 96 | 100 |
  Treatment - Week 102: number analyzed (Participants) | 11 | 0
  Treatment - Week 102 | 84.6 |
  Treatment - Week 108: number analyzed (Participants) | 10 | 0
  Treatment - Week 108 | 100 |
  Treatment - Week 114: number analyzed (Participants) | 5 | 0
  Treatment - Week 114 | 83.3 |
  Treatment - Week 120: number analyzed (Participants) | 4 | 0
  Treatment - Week 120 | 80.0 |
  Treatment - Week 126: number analyzed (Participants) | 3 | 0
  Treatment - Week 126 | 100 |
  Treatment - Week 132: number analyzed (Participants) | 1 | 0
  Treatment - Week 132 | 100 |
  Treatment - Week 138: number analyzed (Participants) | 1 | 0
  Treatment - Week 138 | 100 |

17. Secondary Outcome: Compliance of European Quality of Life (EuroQoL) 5 Dimension 5 Levels (EQ-5D-5L) Questionnaire Over Time
Description: Percentage of participants who filled out an ED-5D-5L questionnaire at a visit. EQ-5D-5L: A generic preference-based health utility measure that provides a single index value for health status. The instrument consists of two parts. The first part, health-state classification, contains five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Time Frame: Baseline through Week 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 72 | 35
percentage of participants
  Treatment - Week 0 | 88.9 | 82.9
  Treatment - Week 3: number analyzed (Participants) | 67 | 33
  Treatment - Week 3 | 86.6 | 78.8
  Treatment - Week 6: number analyzed (Participants) | 62 | 29
  Treatment - Week 6 | 91.9 | 58.6
  Treatment - Week 12: number analyzed (Participants) | 53 | 10
  Treatment - Week 12 | 86.8 | 80
  Treatment - Week 18: number analyzed (Participants) | 43 | 6
  Treatment - Week 18 | 72.1 | 66.7
  Treatment - Week 24: number analyzed (Participants) | 34 | 3
  Treatment - Week 24 | 82.4 | 100
  Treatment - Week 30: number analyzed (Participants) | 25 | 3
  Treatment - Week 30 | 80 | 66.7
  Treatment - Week 36: number analyzed (Participants) | 20 | 2
  Treatment - Week 36 | 80 | 50
  Treatment - Week 42: number analyzed (Participants) | 12 | 2
  Treatment - Week 42 | 91.7 | 50
  Treatment - Week 48: number analyzed (Participants) | 8 | 1
  Treatment - Week 48 | 62.5 | 0
  Treatment - Week 54: number analyzed (Participants) | 3 | 0
  Treatment - Week 54 | 100 |
  Treatment - Week 60: number analyzed (Participants) | 2 | 0
  Treatment - Week 60 | 50 |

18. Secondary Outcome: Time to Deterioration (TTD) in Lung Cancer Symptoms Using EORTC QLQ-LC13 Score for ITT Population
Description: TTD in the overall population is defined as time from randomization to the earliest time with a ≥10-point increase from baseline for symptoms domains (or decrease for functioning domains from baseline for cough, dyspnea [single item and multi-item scales] chest pain [single item], pain in arm/shoulder and fatigue as measured by the EORTC QLQ-LC13.
Time Frame: Baseline through study end (up to 33 months)
Population: ITT population included all participants randomized in the study, irrespective of whether or not they received study drug. Number analyzed indicates number of participants evaluated for specified categories.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
months
  Coughing score | 18.1 [7.2 to NA] — The upper limit of CI was not reached due to an insufficient number of participants with the event. | 16.6 [3.3 to 16.6]
  Dyspnoea score | 4.1 [1.4 to 11.3] | 3.3 [1.0 to NA] — The upper limit of CI was not reached due to an insufficient number of participants with the event.
  Pain in chest score | NA [11.1 to NA] — The median and upper limit of CI was not reached due to less number of participants with the event. | NA [1.6 to NA] — The median and upper limit of CI was not reached due to less number of participants with the event.
  Pain in arm or shoulder score | 12.5 [7.4 to NA] — The upper limit of CI was not reached due to less number of participants with the event. | 1.9 [1.6 to NA] — The upper limit of CI was not reached due to less number of participants with the event.

19. Secondary Outcome: Time to Deterioration (TTD) in Lung Cancer Symptoms Using EORTC QLQ-LC13 Score for C-ITT Population
Description: as for outcome 18
Time Frame: Baseline through study end (up to 33 months)
Population: C-ITT included participants in ITT population with CNS metastasis at baseline (as per IRC assessment). Number analyzed indicates number of participants evaluated for specified categories.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 52 | 28
months
  Coughing score | NA [8.3 to NA] — The median and upper limit of CI were not reached due to an insufficient number of participants with the event. | 16.6 [1.2 to 16.6]
  Dyspnoea score | 9.7 [1.5 to 14.4] | 1.4 [0.8 to NA] — The upper limit of CI was not reached due to an insufficient number of participants with the event.
  Pain in chest score | NA [9.7 to NA] — The upper limit of CI was not reached due to less number of participants with the event. | NA [1.4 to NA] — The median and upper limit of CI was not reached due to less number of participants with the event.
  Pain in arm or shoulder score | 11.1 [4.1 to NA] — The upper limit of CI was not reached due to less number of participants with the event. | 1.7 [0.9 to NA] — The upper limit of CI was not reached due to less number of participants with the event.

20. Secondary Outcome: Time to Deterioration (TTD) in Lung Cancer Symptoms Using EORTC QLQ-LC30 Score for ITT Population
Description: TTD in the overall population is defined as time from randomization to the earliest time with a ≥10-point increase from baseline for symptoms domains (or decrease for functioning domains from baseline for cough, dyspnea [single item and multi-item scales] chest pain [single item], pain in arm/shoulder and fatigue as measured by the EORTC QLQ-C30.
Time Frame: Baseline through study end (up to 33 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
months
  Dyspnoea score | 13.3 [2.9 to NA] — The upper limit of CI was not reached due to an insufficient number of participants with the event. | 8.3 [1.2 to 8.3]
  Fatigue score | 5.6 [1.4 to NA] — The upper limit of CI was not reached due to an insufficient number of participants with the event. | 1.2 [0.8 to NA] — The upper limit of CI was not reached due to an insufficient number of participants with the event.

21. Secondary Outcome: Time to Deterioration (TTD) in Lung Cancer Symptoms Using EORTC QLQ-LC30 Score for C-ITT Population
Description: as for outcome 20
Time Frame: Baseline through study end (up to 33 months)
Population: C-ITT included participants in ITT population with CNS metastasis at baseline (as per IRC assessment).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 52 | 26
months
  Dyspnoea score | 16.6 [2.9 to NA] — The upper limit of CI was not reached due to an insufficient number of participants with the event. | 8.3 [1.0 to 8.3]
  Fatigue score | 14.4 [2.6 to NA] — The upper limit of CI was not reached due to less number of participants with the event. | 1.0 [0.8 to NA] — The upper limit of CI was not reached due to less number of participants with the event.

22. Secondary Outcome: TTD in Composite of Three Symptoms (Cough, Dyspnea, and Chest Pain) Using EORTC QLQ-LC13 Score for C-ITT Population
Description: TTD for a composite of three symptoms (cough, dyspnea, chest pain) in the overall population is defined as time from randomization to the earliest time with a ≥10-point increase from baseline for any component of the composite of the three following symptoms [cough, dyspnea [multi-item subscales QLQ-LC13] and chest pain]) as measured by the EORTC QLQ-LC13.
Time Frame: Baseline through study end (up to 33 months)
Population: C-ITT included participants in ITT population with CNS metastasis at baseline (as per IRC assessment).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 52 | 28
months | 2.8 [0.9 to 5.6] | 1.4 [0.8 to NA] — The upper CT limit could not be estimated due to an insufficient number of participants with the event

23. Secondary Outcome: TTD in Composite of Three Symptoms (Cough, Dyspnea, and Chest Pain) Using EORTC QLQ-LC13 Score for ITT Population
Description: as for outcome 22
Time Frame: Baseline through study end (up to 33 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 79 | 40
months | 1.4 [0.9 to 4.2] | 1.4 [0.9 to 4.2]

24. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline through study end (up to 33 months)
Population: Safety (SAF) population included all participants who received at least one dose of any study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
Number analyzed (Participants) | 77 | 37
Percentage of Participants | 89.6 | 89.2

ADVERSE EVENTS:
Time Frame: Approximately 15 months
Description: SAF population included all participants who received at least one dose of any study drug.
Arm/Group | Experimental: Alectinib | Active Comparator: Premetrexed/Docetaxel
All-Cause Mortality (participants affected / at risk) | 26/77 | 4/37
Serious Adverse Events (participants affected / at risk) | 20/77 | 7/37
Other Adverse Events (participants affected / at risk) | 57/77 | 31/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Alectinib (N=77) | Active Comparator: Premetrexed/Docetaxel (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Abscess jaw (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar ataxia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
H1N1 Influenza (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Death (General disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Alectinib (N=77) | Active Comparator: Premetrexed/Docetaxel (N=37)
Anaemia (Blood and lymphatic system disorders) | 12 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 16 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 3 | 6
Vomiting (Gastrointestinal disorders) | 3 | 2
Asthenia (General disorders) | 9 | 6
Fatigue (General disorders) | 5 | 9
Oedema peripheral (General disorders) | 11 | 2
Pyrexia (General disorders) | 3 | 3
Blood bilirubin increased (Investigations) | 6 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 5 | 3
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 8
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 5 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 2
Bronchitis (Infections and infestations) | 5 | 1
Nasopharyngitis (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 6 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 1
Blood Creatinine Increased (Investigations) | 5 | 0
Electrocardiogram QT Prolonged (Investigations) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT02604342/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT02604342/SAP_003.pdf